CLINICAL TRIAL: NCT02807779
Title: Intima Versus Adventitia Drug Delivery to Elucidate Mechanisms of Restenosis: Magnetic Resonance Imaging
Acronym: INVADER_MRI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Washington (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15-17251; 1R01HL128816-01 (NIH)
Record Dates: First submitted 2016-04-01; First posted 2016-06-21 (Estimated); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Peripheral Artery Disease; Vascular Disease; Critical Limb Ischemia
Keywords: angioplasty; peripheral artery disease; peripheral vascular disease; atherosclerosis; balloon angioplasty; dexamethasone; drug coated balloon; paclitaxel; walking; claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Vascular Diseases; Chronic Limb-Threatening Ischemia; Peripheral Vascular Diseases; Atherosclerosis; Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Dexamethasone (Experimental): Participants randomized to the Dexamethasone group will receive dexamethasone infusion to the adventitia of the artery following plain-old-balloon-angioplasty (POBA).
  Interventions: Drug: Dexamethasone infusion
- Drug Coated Balloon (Active Comparator): Participants randomized to the Drug Coated Balloon (DCB) group will not receive dexamethasone infusion to the adventitia of the artery following (POBA). They will receive additional angioplasty with a paclitaxel coated balloon.
  Interventions: Device: Drug coated balloon
- Plain Balloon Angioplasty (Active Comparator): Participants randomized to the Plain Balloon Angioplasty will receive balloon angioplasty (POBA) only. They will not receive a dexamethasone infusion to the adventitia or paclitaxel.
  Interventions: Device: Plain balloon angioplasty

INTERVENTIONS:
Drug: Dexamethasone infusion — Participants will receive dexamethasone infusion following plain balloon angioplasty
  Other Names: microinfusion catheter
  Arms: Dexamethasone
Device: Drug coated balloon — Participants will receive angioplasty with a drug-coated balloon following plain balloon angioplasty
  Arms: Drug Coated Balloon
Device: Plain balloon angioplasty — Participants will receive plain balloon angioplasty only
  Arms: Plain Balloon Angioplasty

SUMMARY:
This is a prospective, multicenter, randomized trial to determine the mechanisms of vascular healing. The study will evaluate subjects with peripheral artery disease (PAD) who require an endovascular intervention of the femoro-popliteal (SFA) artery to restore blood flow to the leg.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) affects at least 12 million Americans annually with more than half a million patients undergoing an endovascular or surgical revascularization procedure in order to treat the disease. Unfortunately, about two-thirds of patients still have blockages in the leg arteries, even after these procedures.

Advances in Magnetic resonance imaging (MRI) offer promise for understanding the mechanism of failure through insights into vessel wall composition, remodeling, and inflammation. Restenosis has a known relationship to inflammation. Advances in micro-catheter technologies offer the ability to deliver anti-inflammatory medications such as Dexamethasone (DEX) directly to the adventitia and advances in drug delivery on balloon surfaces to deliver paclitaxel to the intima of the artery.

This study aims to investigate if patient-specific parameters affect angioplasty outcomes, if DEX has a biological effect on the vessel wall, and if this effect is through the reduction of inflammation.

In response to an FDA issued "Letter to Healthcare Providers" dated August 9, 2019 that reported the "relative risk for increased mortality at 5 years was 1.57 (95% confidence interval 1.16 - 2.13), which corresponds to a 57% relative increase in mortality in patients treated with paclitaxel-coated devices," participant enrollment in the paclitaxel drug coated balloon arm was stopped and a plain balloon angioplasty arm was added to the protocol.

ELIGIBILITY:
Inclusion Criteria:

Screening:

1. Male or non-pregnant female ≥ 35 years of age
2. Atherosclerotic, infrainguinal PAD
3. Rutherford Clinical Category 2-6
4. Stenosis detected by radiology that in the clinician's opinion is the reason for the PAD symptoms
5. Patient is willing to provide informed consent and comply with the required follow up visits, testing schedule, and medication regimen
6. Estimated Glomerular Filtration Rate (eGFR) ≥ 30 and/or threshold established by the local Institutional Review Board or Committee of Human Research

Procedural Criteria:

1. De novo atherosclerotic lesion qualifying for angioplasty
2. A patent artery proximal to the index lesion. Concomitant inflow procedures, including open femoral artery endarterectomy and/or stenting of the iliac arteries, are permissible.
3. >50% diameter stenosis of the superficial femoral artery and/or popliteal artery (between the profunda and tibioperoneal trunk)
4. Reference vessel diameter ≥3 mm and ≤ 8mm
5. Successful wire crossing of lesion
6. Successful angioplasty of the index lesion or part of the index lesion, defined as ≤30% residual lumen stenosis compared with adjacent non-diseased lumen diameter, without flow-limiting dissection

Exclusion Criteria:

Screening Criteria:

1. Any contraindication to receiving an MRI
2. Pregnant, nursing, or planning on becoming pregnant in < 2yrs
3. Life expectancy of < 1 yr
4. History of solid organ transplantation
5. Patient actively participating in another investigational device or drug study
6. History of hemorrhagic stroke within 3 months of index procedure
7. Previous or planned surgical or interventional procedure within 30 days of index procedure
8. Chronic renal insufficiency with eGFR < 30
9. Prior bypass surgery, stenting, atherectomy or angioplasty of the index lesion
10. Inability to take required study medications
11. Contra-indication or known hypersensitivity to dexamethasone sodium phosphate, contrast media, gadolinium, aspirin or Plavix
12. Systemic fungal infection
13. Acute limb ischemia
14. Prior participation of the index limb in the current study (contralateral treatment is allowed)
15. Patient is being treated with long-term steroids (not including treatment of a bronchial condition with inhaled steroids)

Procedural Criteria:

1. Index lesions extending into the tibial trifurcation or above the profunda. Note: the outflow tibial artery can be treated concomitantly. Similarly, the common femoral artery can be treated concomitantly, either with open endarterectomy and patch angioplasty or with endovascular methods. However, the index lesion cannot be contiguous with either the common femoral artery or the tibial trifurcation.
2. Circumferential calcification at index lesion, which in the judgment of the investigator would prevent penetration of the Micro-Infusion catheter needle through the vessel wall
3. Inadequate distal outflow defined as no patent tibial arteries (>50% stenosis). The outflow vessel can be established at the time of primary treatment
4. Use of adjunctive therapies other than angioplasty. Chocolate balloons and/or scoring balloons are allowed, if used below reference diameter.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren Gasper, MD, Principal Investigator — San Francisco VA Medical Center; David Saloner, PhD, Principal Investigator — San Francisco VA Medical Center
Locations (2):
- United States (2):
  - San Francisco VA Medical Center, San Francisco, California
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 33 enrolled participants, 20 met inclusion criteria and were randomized to treatment.
Groups:
- Dexamethasone: Participants received dexamethasone infusion to the adventitia of the treated artery (1.6mg per cm of artery) following plain-old-balloon-angioplasty (POBA).
  Dexamethasone infusion: Dexamethasone infusion to the artery adventitia (1.6mg per cm of artery) following plain balloon angioplasty
- Drug-Coated Balloon: Participants received additional angioplasty with a paclitaxel drug-coated balloon (DCB) of the treated artery following plain-old-balloon-angioplasty (POBA).
  Drug-coated balloon: Angioplasty with a paclitaxel drug-coated balloon following plain balloon angioplasty
- Plain Balloon Angioplasty: Participants received plain-old-ballon-angioplasty (POBA) only.
  Plain balloon angioplasty: Participants will receive plain balloon angioplasty only
Period: Overall Study
Arm/Group | Dexamethasone | Drug-Coated Balloon | Plain Balloon Angioplasty
Started | 10 | 9 | 1
Completed | 6 | 8 | 0
Not Completed | 4 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 1
Not completed — Death | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone | Drug-Coated Balloon | Plain Balloon Angioplasty | Total
Number analyzed (Participants) | 10 | 9 | 1 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (7.5) | 67.6 (9.9) | 76 (0) | 67.7 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1
  Male | 10 | 8 | 1 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 9 | 1 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 0 | 4
  White | 9 | 6 | 1 | 16
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Hypertension [Count of Participants; unit: Participants] | 10 | 8 | 1 | 19
Hyperlipidemia [Count of Participants; unit: Participants] | 9 | 6 | 0 | 15
Diabetes mellitus [Count of Participants; unit: Participants] | 5 | 3 | 0 | 8
Coronary artery disease [Count of Participants; unit: Participants] | 6 | 2 | 1 | 9
Rutherford category [Count of Participants; unit: Participants] — Rutherford category 1-3 refer to intermittent claudication, less severe presentations of peripheral artery disease Rutherford category 4 refers to ischemic rest pain, a severe presentation of peripheral artery disease Rutherford category 5 refers to ischemic wounds, a severe presentation of peripheral artery disease
  Participants
    Rutherford category 1 | 0 | 0 | 0 | 0
    Rutherford category 2 | 2 | 1 | 0 | 3
    Rutherford category 3 | 7 | 8 | 1 | 16
    Rutherford category 4 | 0 | 0 | 0 | 0
    Rutherford category 5 | 1 | 0 | 0 | 1
White blood cell count [Mean (Standard Deviation); unit: 10^9 cells/L] | 8.6 (1.8) | 7.9 (2.2) | 8 (0) | 8.2 (1.9)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 12.3 (1.6) | 12.9 (1.1) | 14.6 (0) | 12.7 (1.4)
Hematocrit [Mean (Standard Deviation); unit: percentage of hematocrit] | 37.5 (4.8) | 38.8 (3.2) | 43.2 (0) | 38.4 (4.1)
Platelet count [Mean (Standard Deviation); unit: 10^9 platelets/L] | 225.1 (62.3) | 244.5 (62.9) | 157 (0) | 229.9 (62.3)
C-Reactive Protein (CRP) [Median (Inter-Quartile Range); unit: mg/L] | 3.5 [1.6 to 12.3] | 2.0 [1.0 to 3.6] | .33 [.33 to .33] | 2.1 [.96 to 6.4]
Monocyte Chemotactic Protein 1 (MCP-1) [Mean (Standard Deviation); unit: pg/mL] | 72.6 (21.5) | 77.1 (19.6) | 62.0 (0) | 73.9 (19.8)
Interleukin 1 Beta (IL-1beta) [Median (Inter-Quartile Range); unit: pg/mL] | 0.19 [0.11 to 0.91] | 0.17 [0.10 to 0.24] | 0 [0 to 0] | 0.19 [0.11 to 0.24]

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent Wall Volume (PWV)
Description: The change in percent wall volume (PWV) of the treated segment between the postoperative and 12 month time points as measured by MRI
Time Frame: From Post-Operative Day One to 12 Months
Population: No data was collected for the Plain Balloon Angioplasty group
Measure: Mean (Standard Deviation); unit: Percent Wall Volume
Arm/Group | Dexamethasone | Drug-Coated Balloon | Plain Balloon Angioplasty
Number analyzed (Participants) | 5 | 4 | 0
Percent Wall Volume | 12.3 (11.6) | 3.9 (4.3) |
Statistical Analysis 1: Comparison: Dexamethasone vs Drug-Coated Balloon; Power calculations were performed based on an expected reproducibility variance of 8% and an effect size of 7% was assumed based on data from pilot studies. It was estimated that 22 subjects/treatment assignment were needed to detect a 7% difference in PWV at a power level of 80%. Assigning a 20% attrition rate due to loss to follow up or index lesion revascularization, the goal enrollment was 27 subjects per arm. No subjects in the plain balloon angioplasty group had MRI data for analysis; Test type: Superiority; p = 0.22, t-test, 2 sided — Threshold for statistical significance was p=0.05

2. Secondary Outcome: Change in Wall Volume (WV) Without a Change in Total Vessel Volume (TVV)
Description: The change in wall volume (WV) without change in total vessel volume (TVV) of the treated segment between the postoperative and 12 month time points as measured by MRI
Time Frame: From Post-Operative Day One to 12 Months
Population: No data was collected for the Plain Balloon Angioplasty group
Measure: Mean (Standard Deviation); unit: mm*3
Arm/Group | Dexamethasone | Drug-Coated Balloon | Plain Balloon Angioplasty
Number analyzed (Participants) | 5 | 4 | 0
mm*3 | 28.7 (78.5) | 4.5 (66.6) |
Statistical Analysis 1: Comparison: Dexamethasone vs Drug-Coated Balloon; No subjects in the plain balloon angioplasty group had MRI data for analysis; Test type: Superiority; p = 0.64, t-test, 2 sided — Threshold for statistical significance was p=0.05

3. Secondary Outcome: Change in Perioperative Inflammatory Profile (MCP-1)
Description: The serum concentration of monocyte chemoattractant protein-1 (MCP-1) between postprocedure day 1 and 12 months postprocedure. Reported as the area under the curve (AUC) of the MCP-1 concentration (postprocedure day 1, 1 month and 12 months)
Time Frame: From Post-Operative Day One to 12 Months
Population: No data was collected for the Plain Balloon Angioplasty group
Measure: Mean (Standard Deviation); unit: pg*d/mL
Arm/Group | Dexamethasone | Drug-Coated Balloon | Plain Balloon Angioplasty
Number analyzed (Participants) | 6 | 4 | 0
pg*d/mL | 27933 (3267) | 277745 (4000) |
Statistical Analysis 1: Comparison: Dexamethasone vs Drug-Coated Balloon; No subjects in the plain balloon angioplasty group had complete MCP-1 data for analysis; Test type: Superiority; p = 0.95, t-test, 2 sided — Threshold for statistical significance was p=0.05

4. Secondary Outcome: Change in Perioperative Inflammatory Profile (CRP)
Description: The serum concentration of C-reactive protein (CRP) between postprocedure day 1 and 12 months postprocedure. Reported as the area under the curve (AUC) of the CRP concentration (postprocedure day 1, 1 month and 12 months).
Time Frame: From Post-Operative Day One to 12 Months
Population: No data was collected for the Plain Balloon Angioplasty group
Measure: Mean (Standard Deviation); unit: mg*d/L
Arm/Group | Dexamethasone | Drug-Coated Balloon | Plain Balloon Angioplasty
Number analyzed (Participants) | 6 | 4 | 0
mg*d/L | 1721 (1171) | 1863 (1475) |
Statistical Analysis 1: Comparison: Dexamethasone vs Drug-Coated Balloon; No subjects in the plain balloon angioplasty group had complete CRP data for analysis; Test type: Superiority; p = 0.88, t-test, 2 sided — Threshold for statistical significance was p=0.05

5. Secondary Outcome: Change in Perioperative Inflammatory Profile (IL-1beta)
Description: The serum concentration of interleukin-1beta (IL-1beta) between postprocedure day 1 and 12 months postprocedure. Reported as the area under the curve (AUC) of the IL-1beta concentration (postprocedure day 1, 1 month and 12 months).
Time Frame: From Post-Operative Day One to 12 Months
Population: No subject had measurable serum IL-1beta at the 12month timepoint
Arm/Group | Dexamethasone | Drug-Coated Balloon | Plain Balloon Angioplasty
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change in Transfer Constant (Ktrans)
Description: The change in adventitial transfer constant (Ktrans) of the treated segment between the postoperative and 6 month time points as measured by dynamic contrast enhanced MRI
Time Frame: From 1 Month to 6 Months
Population: No data was collected for the Plain Balloon Angioplasty group
Measure: Mean (Standard Deviation); unit: min^-1
Arm/Group | Dexamethasone | Drug-Coated Balloon | Plain Balloon Angioplasty
Number analyzed (Participants) | 6 | 4 | 0
min^-1 | -0.0002 (0.003) | -0.0067 (0.006) |
Statistical Analysis 1: Comparison: Dexamethasone vs Drug-Coated Balloon; No subjects in the plain balloon angioplasty group had MRI data for analysis; Test type: Superiority; p = .055, t-test, 2 sided — Threshold for statistical significance was p=0.05

7. Secondary Outcome: Change in Lumen Volume (LV) Relative to Total Vessel Volume (TVV)
Description: The change in lumen volume (LV) relative to total vessel volume (TVV) of the treated segment between the postoperative and 12 month time points as measured by MRI
Time Frame: From Post-Operative Day One to 12 Months
Population: No data was collected for the Plain Balloon Angioplasty group
Measure: Mean (Standard Deviation); unit: mm*3
Arm/Group | Dexamethasone | Drug-Coated Balloon | Plain Balloon Angioplasty
Number analyzed (Participants) | 5 | 4 | 0
mm*3 | -12.3 (11.6) | -3.88 (4.28) |
Statistical Analysis 1: Comparison: Dexamethasone vs Drug-Coated Balloon; No subjects in the plain balloon angioplasty group had MRI data for analysis; Test type: Superiority; p = .22, t-test, 2 sided — Threshold for statistical significance was p=0.05

8. Secondary Outcome: Percentage of Subjects With Clinically Significant Restenosis That Undergo Reintervention of Greater Than or Equal to 75% of the Treated Segment
Description: Percentage of subjects with clinically significant restenosis that undergo reintervention of greater than or equal to 75% of the treated segment by the 12 month timepoint.
Time Frame: From Post-Operative Day One to 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone | Drug-Coated Balloon | Plain Balloon Angioplasty
Number analyzed (Participants) | 10 | 9 | 1
Participants | 4 | 4 | 1
Statistical Analysis 1: Comparison: Dexamethasone vs Drug-Coated Balloon vs Plain Balloon Angioplasty; Test type: Superiority; p = 0.81, Fisher Exact — Threshold for statistical significance was p=0.05

9. Other Pre Specified Outcome: Extended Clinical Adverse Events Monitoring
Description: Participant monitoring for clinical adverse events
Time Frame: From Post-Operative Day One to 36 Months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 36 months
Description: Adverse Event data collection for 36 months after index procedure
Arm/Group | Dexamethasone | Drug-Coated Balloon | Plain Balloon Angioplasty
All-Cause Mortality (participants affected / at risk) | 1/10 | 1/9 | 0/1
Serious Adverse Events (participants affected / at risk) | 7/10 | 7/9 | 1/1
Other Adverse Events (participants affected / at risk) | 1/10 | 1/9 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone (N=10) | Drug-Coated Balloon (N=9) | Plain Balloon Angioplasty (N=1)
Death (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Reintervention requiring hospitalization (Vascular disorders) | 5 (10) | 6 (7) | 1 (2) — Repeat procedure on the arteries of the treated (index) or non-treated (non-index) leg requiring hospitalization
COVID pneumonia requiring hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0
Acute heart failure requiring admission (Cardiac disorders) | 1 (1) | 0 | 0
Arterial access site pseudoaneurysm requiring operation (Vascular disorders) | 0 | 0 | 1 (1)
Unstable angina requiring coronary revascularization (Cardiac disorders) | 1 (1) | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone (N=10) | Drug-Coated Balloon (N=9) | Plain Balloon Angioplasty (N=1)
Pacemaker placement (Cardiac disorders) | 1 (1) | 0 | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 1 | 0 — Urinary tract infection leading to ER visit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT02807779/Prot_SAP_001.pdf